CLINICAL TRIAL: NCT01548079
Title: Effects of Ursodeoxycholic Acid on Hepatobiliary Detoxification/Elimination Mechanisms and Hepatic Fatty Acid/Triglyceride Metabolism in Morbidly Obese Patients.
Brief Title: Ursodeoxycholic Acid in Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Hanns-Ulrich Marschall, Professor, senior consultant, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UDCAINBS
Record Dates: First submitted 2012-02-22; First posted 2012-03-08 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Non-alcoholic Fatty Liver Disease; Morbid Obesity
Keywords: ursodeoxycholic acid; fatty liver disease; morbid obesity; bariatric surgery; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity, Morbid | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Untreated controls
- Ursodeoxycholic acid (Active Comparator): Oral ursodeoxycholic acid 20 mg/kg/day in three weeks
  Interventions: Drug: Ursodeoxycholic Acid (UDCA)

INTERVENTIONS:
Drug: Ursodeoxycholic Acid (UDCA) — 20mg/kg/day UDCA in three weeks
  Arms: Ursodeoxycholic acid

SUMMARY:
In an open-label trial, 20 otherwise healthy morbidly obese patients scheduled for bariatric surgery will be administered 20 mg/kg/day ursodeoxycholic acid for three weeks until the day before surgery. The maximum dose will be 3 g/day. Twenty other patients will serve as controls. Serum from days 1 and 21 will be analyzed for routine liver tests, bile acids, a complete lipid profile including FA and in addition for 7α-hydroxy-4-cholesten-3-one and fibroblast growth factor 19 (FGF-19), markers for bile acid synthesis its intestinal stimulation. For the evaluation of insulin resistance and possible pre-diabetes, plasma will be taken for the estimation of homeostasis model assessment (HOMA) index and oral glucose tolerance test (OGTT) will be performed at days 1 and 21. At surgery, a liver biopsy (0.5-1 g) and a white adipose tissue (WAT) specimen (1 cm2) will be taken and immediately frozen in liquid nitrogen for messenger ribonucleic acid (mRNA) and protein preparation for quantitative real-time polymerase chain reaction (RT-PCR) and Western analysis, respectively, histopathological Non-alcoholic fatty liver disease (NAFLD) grading, and measuring of hepatic and white adipose tissue (WAT) lipase activity. In all patients at randomization, abdominal ultrasound will be performed for the detection of NAFLD and gallstones and a blood sample will be taken for the analysis of polymorphisms of hepatic lipid synthesis, storage, fatty acid (FA) oxidation and export genes. Six month after operation, HOMA, OGTT and abdominal ultrasound will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 35 kg/m2
* Patients eligible to bariatric surgery
* Patients should have given their written consent to participate in this study

Exclusion Criteria:

* Chronic liver disease other than NAFLD (viral hepatitis, autoimmune liver disease, hemochromatosis, homozygous alpha1-antitrypsin deficiency and Wilson disease)
* Partial ileal bypass
* Inflammatory bowel disease
* Uncontrolled diabetes mellitus (fasting blood glucose > 6.7 mmol/L), hypothyroidism or hyperthyroidism, or other significant endocrine disease.
* A subject who is euthyroid on a stable replacement dose of thyroid hormone is acceptable provided the TSH is within normal range.
* Other serious disease
* Known hypersensitivity to ursodeoxycholic acid
* Patients who will not comply with the protocol.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Changes in regulators of lipid turnover | Baseline and 3 weeks
  Trial objectives are to determine whether (i) Hepatic and/or visceral white adipose tissue (WAT) lipase activity determines fatty acid (FA) release/balance from lipid triglyceride (TG) droplets and FA-mediated lipotoxicity in NAFLD; differences in hepatic and/or WAT activity could explain individual susceptibility to pure NAFL versus NASH (ii) UDCA (20 mg/kg/day) improves insulin resistance in patients with NAFLD (iii) UDCA improves hepatobiliary transporter expression in NAFLD

SECONDARY OUTCOMES:
Changes in serum bile acids and lipids | Baseline and 3 weeks
  * relative changes in hepatic basolateral transport proteins MRP3, MRP4, OATP, SLC21A1
  * relative changes in m RNA expression levels of BAAT; CYP3A4, CYP7A1, CYP27, CYP8B1, UGT1A1, UGT2B4, UGT2B7, SULT2A1, HNF-4α, PXR/NR1I2, RXR/NR1B1; PERK, XBP-1, SREBP-1c; TNF-α, IL-6, IL-10, MCP-1, CxCl-1
  * relative change in serum bile acids
  * relative change in plasma 7α-hydroxy-4-cholesten-3-one and FGF-19
  * relative changes in total cholesterol, LDL-C, HDL-C, Apo A1, Apo B, in Lp(A)

CONTACTS AND LOCATIONS:
Overall Officials: Hanns-Ulrich Marschall, MD, PhD, Principal Investigator — Sahlgrenska Academy and University Hospital, Institute of Medicine, Dept. of Internal Medicine, University of Gothenburg, S-41345 Gothenburg

REFERENCES:
- [Derived] Mueller M, Castro RE, Thorell A, Marschall HU, Auer N, Herac M, Rodrigues CMP, Trauner M. Ursodeoxycholic acid: Effects on hepatic unfolded protein response, apoptosis and oxidative stress in morbidly obese patients. Liver Int. 2018 Mar;38(3):523-531. doi: 10.1111/liv.13562. Epub 2017 Sep 18. PMID 28853202